CLINICAL TRIAL: NCT05142813
Title: A Cohort Study to Evaluate Biomarkers as Indicator for the Infectious Source of Sepsis Through a Blood Test
Brief Title: A Blood Test to Diagnose Sepsis in Symptomatic Adults and Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: mProbe Inc. (Industry)
Collaborators: The Second Afliated Hospital of Southern University of Science and Technology (Unknown)
Responsible Party: Principal Investigator, Jia Huang, Principal Investigator, mProbe Inc.
Other Study IDs: Sepsis_001
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Infections; Sepsis; SIRS
Keywords: Acute infection; Fever without source; Viral infection
MeSH Terms: conditions — Infections; Sepsis; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Blood specimen collection — Diagnostic Test: Blood specimen collection Study samples must be collected within before treatment with antibiotics or antivirals.

SUMMARY:
A case-control cohort study to develop and validate the performance of a whole blood gene expression test to distinguish sepsis infection from uninfected systemic inflammatory response syndrome cases in symptomatic adults and children without comorbidities.

DETAILED DESCRIPTION:
The purpose of this prospective, non-interventional study is to develop and validate a blood gene expression test for diagnosing the cause of sepsis in adults and children with symptoms of infection.

Sepsis affects 31.5 million people globally leading to 5.3 million deaths each year. Sepsis is particularly harmful to immunodeficient patients undergoing cancer therapy with 3.7 percent to 6.4 percent of cancer patients diagnosed with sepsis in the US in their first year after cancer diagnosis. Current tests to diagnose the infectious cause of sepsis rely on blood cultures which takes 24-48 hours to complete; leading to delays in early treatment critical to reduce the risk of developing sepsis shock and possibly death. In addition, around 50 percent of severe sepsis cases are culture negative, confounded acute infections not detected in the blood, by viral infection or uninfected patients exhibiting systemic inflammatory response syndrome (SIRS). Since sepsis often progresses to sepsis shock within 72 hours, suspected sepsis cases are usually immediately treated with antibiotics until results from testing distinguish the cause of symptoms. This leads to the over-use of antibiotics and delays appropriate treatment for those without bacterial infection or un-infected SIRS.

A quick and accurate diagnostic blood test may enable early discrimination of the cause of sepsis resulting in faster more appropriate treatments and reduced sepsis complications and death.

The study will collect blood samples from participants presenting symptoms of acute infection, without co-morbidities and follow symptom severity and mortality for 28 days.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Clinical suspicion of an acute infectious disease
* Presence of at least ONE of the following:

  1. Temperature ≥ 38°C or Temperature ≤ 36°C
  2. Heart rate > 90 bpm
  3. Respiratory rate > 20/min
  4. Self reported fever/chills
* Symptom duration ≤ 7 days

Exclusion Criteria:

* Received antibiotics or antivirals in the past 2 weeks.
* Previous infection in previous 2 weeks
* Primary or secondary immunodeficiency
* Proven or suspected HIV, hepatitis B or hepatitis C infection
* Current immune-suppressive or immune-modulating treatment
* Active hematological malignancy
* Other illnesses that affect life expectancy

Ages: 90 Days to 85 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants 90 days of age and older that visit the hospital or emergency department with a suspected acute infection.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of underlying cause of sepsis infection | 1 month
  The sensitivity and specificity of the assay in differentiating bacterial from viral infection.

SECONDARY OUTCOMES:
Diagnosis of underlying cause of acute infection symptoms | 1 month
  The sensitivity and specificity of the assay in differentiating infectious and non-infectious disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Huang, Principal Investigator — The Second Afliated Hospital of Southern University of Science and Technology